CLINICAL TRIAL: NCT04148482
Title: PREMIER: PREvention of Metabolic Illness Through prEcision nutRition
Acronym: PREMIER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); NORCH (Nutrition Obesity Research Center at Harvard) (Unknown); Boston Area Diabetes Endocrinology Research Center (Unknown)
Responsible Party: Principal Investigator, Sara Cromer, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 2019P002638; P30DK040561 (NIH)
Record Dates: First submitted 2019-10-18; First posted 2019-11-01 (Actual); Results first posted 2025-06-08 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Obesity; Type 2 Diabetes; Metabolic Syndrome; Diet Habit; Nutritional and Metabolic Disease; Food Preferences
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Metabolic Syndrome; Feeding Behavior; Metabolic Diseases; Food Preferences | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: This is a recall-by-genotype study
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genotype of interest group (Active Comparator): Individuals with desired genetic susceptibility will receive a standardized and an election meal in a full-day clinic visit.
  Interventions: Other: Dietary intervention
- Control (Placebo Comparator): Individuals without genotype of interest (i.e., carrying the opposite genotype) will receive a standardized and an election meal in a full-day clinic visit.
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention — To investigate whether individuals with divergent genetic susceptibility have different food preferences and have differential post-prandial glycemic and metabolomics responses to a standardized or an election meal.

SUMMARY:
Dietary intake is a major driving force behind the escalating obesity and type 2 diabetes epidemics. Large, high-quality clinical trials have shown that close adherence to healthy dietary recommendations significantly reduce the incidence of obesity and type 2 diabetes, especially among people at increased risk. However, large inter-individual variability exists in response to dietary interventions. To inform more effective obesity and type 2 diabetes prevention strategies, it is crucial to better understand the biological, environmental, and social factors that influence how people interact and respond to specific foods.

In a recent large-scale genome-wide association study, our research team has identified 96 genomic regions associated with overall variation in dietary intake. This study provided evidence that inherited molecular differences are likely to impact on food intake (i.e., preference for certain foods) and metabolic homeostasis (i.e., glucose regulation). Connecting knowledge about human genetic variants with information from circulating metabolites can be particularly useful in understanding the mechanisms by which some people experience a detrimental response to specific foods.

The specific objective of the PREMIER study is to carry out an interventional dietary study to measure the response of blood glucose and other biomarkers to a standardized meal, and evaluate the extent to which food choices differ among individuals with distinct genetic susceptibility.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* 21-65 years of age.
* Body mass index (BMI) between 18.5 and 30.0 kg/m2.
* Healthy (free of diagnosed diseases listed in the exclusion criteria).
* Willing to comply with the study intervention.
* Able to provide informed consent

Exclusion Criteria:

* Refuse or are unable to give informed consent to participate in the study.
* Have type I or type II diabetes mellitus or are taking medications for type II diabetes mellitus. Those not on medications but having a capillary glucose level of >126 mg/dL based on fingertip glucose measurements will be excluded.
* Are obese (BMI>30.0kg/m2) or underweight (BMI<18.5kg/m2).
* Have had a heart attack (myocardial infarction) or stroke
* Have had cancer in the last 3 years, excluding skin cancer.
* Have an ongoing inflammatory disease i.e. Rheumatoid arthritis, systemic lupus erythematosus, polymyalgia and other connective tissue diseases.
* History of cirrhosis and/or aspartate aminotransferase (AST) or alanine aminotransferase (ALT) more than 3 times the upper limit of normal (ULN).
* Are currently suffering from acute clinically diagnosed depression.
* Currently taking or intending to take during the study duration any medication known to affect glycemic parameters, such as glucocorticoids or fluoroquinolones.
* Are unable to fast from 9pm the night before the clinic visit until 9am on the clinic day
* Are pregnant or breastfeeding.
* Are participating in another clinical study.
* Are vegan, suffering from an eating disorder or unwilling to eat foods that are part of the study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2024-09-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massacusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Our research team will provide a personalized report containing individual's glycemic responses and potentially other biomarker responses to meals consumed by the end of the study.
Supporting Information: CSR
Time Frame: 6-12 months after finishing the study intervention

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Genotype of Interest Group | Control
Started | 12 | 10
Completed | 12 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Genotype of Interest Group | Control | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 7 | 18
  >=65 years | 1 | 3 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (8.9) | 57.5 (8.3) | 56.2 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 11 | 10 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 12 | 8 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 10 | 22
Glucose at time 0 [Mean (Standard Deviation); unit: mg/dL] | 81.9 (11.7) | 85.6 (8.3) | 83.6 (10.2)

OUTCOME MEASURES:

1. Primary Outcome: Glucose at Times 30min, 60min, 120min, 180min
Description: Measurement of blood glucose at regular intervals.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Genotype of Interest Group | Control
Number analyzed (Participants) | 12 | 10
mg/dL
  30min | 112.9 (19.3) | 119.8 (15.6)
  60min | 94.5 (24.1) | 118.4 (34.3)
  120min | 84.1 (22.5) | 94.1 (10.9)
  180min | 80.8 (12.5) | 81.9 (9.4)

2. Primary Outcome: High-fat Meal Preference
Description: Number of participants with preference for a high-fat meal.
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Genotype of Interest Group | Control
Number analyzed (Participants) | 12 | 10
Participants | 8 | 3

3. Secondary Outcome: Metabolomics by Mass Spectrometry Analysis (Reported as Fold Change in Metabolites From Baseline)
Description: Investigators will perform metabolomic profiling of plasma samples at regular intervals by using both targeted and untargeted approaches on an existing platform that measures ~10,000 metabolites (both polar and non-polar); they will compare their relative concentrations (fold change) by genotype at selected loci before and after the interventions. Metabolomics will be performed using LC-MS techniques in the Clish Laboratory of the Broad Institute of MIT and Harvard (Cambridge, MA). Fold-change in metabolite values (from 0->120, 0->240, and 240->360 minutes) will be statistically analyzed to identify distinct patterns of metabolite change in response to mixed meals by genotype. Examples of metabolomic fold-change readouts are provided below, by genotype - limited examples are provided as fold-change reporting for ~10,000 metabolites, identified and unidentified, at 3 time points would be impracticable.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: fold-change from baseline
Arm/Group | Genotype of Interest Group | Control
Number analyzed (Participants) | 12 | 10
fold-change from baseline
  taurodeoxycholic acid at 120 minutes | 10.4 (8.8) | 4.2 (4.0)
  glycochenodeoxycholic acid at 120 minutes | 6.7 (5.3) | 3.9 (4.5)

4. Other Pre Specified Outcome: Previously Proposed Outcomes: Hunger Perception, Incretin Levels by Immunoassay Kit, Satiety Hormones
Description: Although these outcomes were initially proposed/intended, insufficient funds were available to collect or analyze these measures, and they were not ultimately collected.
Time Frame: baseline, 120min, 240min, 360min
Population: Although these outcomes were initially proposed/intended, insufficient funds were available to collect or analyze these measures, and they were not ultimately collected.
Arm/Group | Genotype of Interest Group | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 8 hours
Arm/Group | Genotype of Interest Group | Control
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 0/12 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-08-15): https://cdn.clinicaltrials.gov/large-docs/82/NCT04148482/Prot_000.pdf
  • Statistical Analysis Plan (2025-04-22): https://cdn.clinicaltrials.gov/large-docs/82/NCT04148482/SAP_001.pdf